CLINICAL TRIAL: NCT05953714
Title: THE EFFECT OF USING CHLORHEXIDINE GLUCONATE AND POVIDONE IODINE SOLUTION ON THE HEALING PROCESS BEFORE A CESAREAN SECTION
Brief Title: CHLORHEXIDINE GLUCONATE AND POVIDONE IODINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Assistant Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHLORHEXIDINE
Record Dates: First submitted 2023-07-03; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Evaluate to Effects of Two Antiseptic Products and Showering
Keywords: Cesarean section; surgical site infection; povidone iodine; chlorhexidine gluconate; patient comfort; healing process
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: They were randomly divided into povidone iodine (PI) group (A) clorhexidine gluconate (CG) group (B) and CG shower (C) operated by two Gynecology and Obstetrics physician. Data from the in house blinding study to avoid bias and follow-up of the women was done for 7 day duration following postnatal to assess postoperative for comfort, pain, wound complications.
Who Masked: Participant
Masking Description: The inclusion criteria included the absence of systemic and chronic disease (thyroid disease, gestational diabetes, gestational hypertension or allergy), no history of previous abdominal surgery, a newborn baby follow-up with no health problems that would hinder the breastfeeding process, 37 gestational weeks of pregnancy and above, pregnant women with a low-risk pregnancy, those with a body mass index between 20 and 30 who were at least a primary school graduate, and who were between 19 to 40 years of age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHLORHEXIDINE GLUCONATE GROUP (Experimental): Section area is cleaned with preoperative application chlorhexidine gluconate
  Interventions: Other: incision side cleaning with antiseptic products
- POVIDONE IODINE GROUP (No Intervention): Section area is cleaned with preoperative application povidone iodine
- CHLORHEXIDINE GLUCONATE SHOWER GROUP (Experimental): Section area is cleaned with preoperative application chlorhexidine gluconate shower
  Interventions: Other: incision side cleaning with antiseptic products

INTERVENTIONS:
Other: incision side cleaning with antiseptic products — A pilot study was conducted with six pregnant women to clarify the use of the data collection tools and the implementation plan during the study process. After that, the data collection forms were finalized. In the 6 operating room, two different solutions (PI and CG) were applied, according to the preference of the physician, to clean the surgical field. The study was carried out by adding a CG shower application to the physician's preferred solution (for a total of 3 groups). Pregnant women who were admitted to the obstetrics clinic were informed about the purpose, scope, duration, and method of the study by one of the researchers. Follow-up of the women was done for 7 day duration following postnatal to assess postoperative for comfort, pain, wound complications by the nurse researcher. At discharge, cultures were taken from the abdominal wounds of the participants
  Arms: CHLORHEXIDINE GLUCONATE GROUP; CHLORHEXIDINE GLUCONATE SHOWER GROUP

SUMMARY:
The study was planned to evaluate the effects of two most commonly used antiseptic products and showering on the healing process, such as wound healing and postoperative maternal comfort in cesarean section. A randomized controlled trial included 102 pregnant women from February and May of 2021. They were randomly divided into povidone iodine (PI) group (A) chlorhexidine gluconate (CG) group (B) and CG shower (C) operated by two Gynecology and Obstetrics physician. Data from the in house blinding study to avoid bias and follow-up of the women was done for 7 day duration following postnatal to assess postoperative for comfort, pain, wound complications.

DETAILED DESCRIPTION:
Purpose and type of research This study was designed as a randomized controlled trial to examine the effect of preoperative use of CG and PI on the postoperative healing process and maternal postpartum comfort.

Hypothesis H1: Cleaning the incision area with a 2% CG solution (containing 70% alcohol) is more effective in the wound healing process than PI.

H2: Taking a shower with a 2% CG solution (containing 70% alcohol) 6 hours before, and cleaning the incision area, is more effective in the wound healing process than PI.

H3: Cleaning the incision area with a 2% CG solution (containing 70% alcohol) produces a higher postpartum comfort level than PI.

H4: Taking a shower 6 hours before with a 2% CG solution (containing 70% alcohol), and cleaning the incision area, produces a higher postpartum comfort level than PI.

Variables in the study include dependent variables: signs of the wound healing process at the incision site (erythema, edema, ecchymosis, discharge, wound dehiscence and pain), and independent variables: a 2% CG (70% alcohol) solution and the application of PI.

Participants This research was carried out in a Turkish research hospital clinic between February and May of 2021. The study sample consisted of all pregnant women (n = 504) who were hospitalized with a planned cesarean section scheduled between the study dates. The study sample consisted of 102 pregnant women who met the inclusion criteria and who agreed to participate in the study after informed consent was obtained. They were randomly divided into groups. The study sample consisted of three groups: 1) those cleaned with povidone-iodine (PI) before the surgical incision, 2) those cleaned with chlorhexidine gluconate (CG) before the surgical incision and 3) those showering with CG six hours before the surgical incision and cleaned with CG before the surgical incision.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized with a planned cesarean section scheduled between the study dates
* volunteer woman

Exclusion Criteria:

* participants who dont meet the inclusion criteria
* labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women who were admitted to the obstetrics clinic were informed about the purpose, scope, duration, and method of the study by one of the researchers.
Enrollment: 102 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
To determine that cleaning the incision site with 2% CG solution (containing 70% alcohol) is more effective than PI in the wound healing process. | 4 months
  To determine that using the Incision site evaluation form (ISEF). This form was used to evaluate erythema, warmth, oedema, discharge and wound opening. The score of form is between 0-3 for each item, and the total score is between 0-15. According to the form, a high score is interpreted as a poor recovery.

SECONDARY OUTCOMES:
To determine that taking a shower with 2% CG solution (containing 70% alcohol) 6 hours before and cleaning the incision site is more effective than PI in the wound healing process. | 4 months
  To determine that using the Incision site evaluation form (ISEF). This form was used to evaluate erythema, warmth, oedema, discharge and wound opening. The score of form is between 0-3 for each item, and the total score is between 0-15. According to the form, a high score is interpreted as a poor recovery.
To determine that cleaning the incision site with 2% CG solution (containing 70% alcohol) provides a higher level of postpartum comfort than PI | 4 months
  The Postpartum Comfort Questionnaire (PPCQ) is a scale that evaluates the physical, psycho-spiritual and sociocultural comfort of mothers who had cesarean and normal births. Physical comfort is defined as psycho-spiritual comfort, the relationship between spirituality and mind, as physiological indicators that can contribute to the healing process, socio-cultural comfort, and relations with family and environment. There are positive and negative items in the five-point Likert-type scale, which consists of thirty-four items, with the lowest possible score being 34 and the highest score being 170. A higher score indicates a higher level of comfort. Comfort status was determined with this questionnaire.
To determine that showering with 2% CG solution (containing 70% alcohol) 6 hours ago and cleaning the incision area provides a higher level of postpartum comfort compared to PI. | 4 months
  The Postpartum Comfort Questionnaire (PPCQ) is a scale that evaluates the physical, psycho-spiritual and sociocultural comfort of mothers who had cesarean and normal births. Physical comfort is defined as psycho-spiritual comfort, the relationship between spirituality and mind, as physiological indicators that can contribute to the healing process, socio-cultural comfort, and relations with family and environment. There are positive and negative items in the five-point Likert-type scale, which consists of thirty-four items, with the lowest possible score being 34 and the highest score being 170. A higher score indicates a higher level of comfort. Comfort status was determined with this questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After our study will be published, we will share our detail information about our study

REFERENCES:
- [Background] Lai YL, Hung CH, Stocker J, Chan TF, Liu Y. Postpartum fatigue, baby-care activities, and maternal-infant attachment of vaginal and cesarean births following rooming-in. Appl Nurs Res. 2015 May;28(2):116-20. doi: 10.1016/j.apnr.2014.08.002. Epub 2014 Oct 23. PMID 25468429
- [Result] Villers MS. Reducing Cesarean Delivery Surgical Site Complications. Obstet Gynecol Clin North Am. 2020 Sep;47(3):429-437. doi: 10.1016/j.ogc.2020.04.006. Epub 2020 Jun 6. PMID 32762928
- [Result] Corcoran S, Jackson V, Coulter-Smith S, Loughrey J, McKenna P, Cafferkey M. Surgical site infection after cesarean section: implementing 3 changes to improve the quality of patient care. Am J Infect Control. 2013 Dec;41(12):1258-63. doi: 10.1016/j.ajic.2013.04.020. Epub 2013 Aug 9. PMID 23938001
- [Result] Charehbili A, Koek MBG, de Mol van Otterloo JCA, Bronkhorst MWGA, van der Zwaal P, Thomassen B, Waasdorp EJ, Govaert JA, Bosman A, van den Bremer J, Ploeg AJ, Putter H, Meijs AP, van de Velde CJH, van Gijn W, Swijnenburg RJ. Cluster-randomized crossover trial of chlorhexidine-alcohol versus iodine-alcohol for prevention of surgical-site infection (SKINFECT trial). BJS Open. 2019 May 20;3(5):617-622. doi: 10.1002/bjs5.50177. eCollection 2019 Oct. PMID 31592513
- [Result] Burke C, Allen R. Complications of Cesarean Birth: Clinical Recommendations for Prevention and Management. MCN Am J Matern Child Nurs. 2020 Mar/Apr;45(2):92-99. doi: 10.1097/NMC.0000000000000598. PMID 31804227
- [Result] Money L, Eyer M, Duncan K. Creating a Surgical Site Infection Prevention Bundle for Patients Undergoing Cesarean Delivery: 1.6 www.aornjournal.org/content/cme. AORN J. 2018 Oct;108(4):372-383. doi: 10.1002/aorn.12371. PMID 30265380
- [Result] Kawakita T, Landy HJ. Surgical site infections after cesarean delivery: epidemiology, prevention and treatment. Matern Health Neonatol Perinatol. 2017 Jul 5;3:12. doi: 10.1186/s40748-017-0051-3. eCollection 2017. PMID 28690864
- [Result] Huang H, Li G, Wang H, He M. Optimal skin antiseptic agents for prevention of surgical site infection in cesarean section: a meta-analysis with trial sequential analysis. J Matern Fetal Neonatal Med. 2018 Dec;31(24):3267-3274. doi: 10.1080/14767058.2017.1368481. Epub 2017 Aug 30. PMID 28817989
- [Result] Stone J, Bianco A, Monro J, Overybey JR, Cadet J, Choi KH, Pena J, Robles BN, Mella MT, Matthews KC, Factor SH. Study To Reduce Infection Prior to Elective Cesarean Deliveries (STRIPES): a randomized clinical trial of chlorhexidine. Am J Obstet Gynecol. 2020 Jul;223(1):113.e1-113.e11. doi: 10.1016/j.ajog.2020.05.021. Epub 2020 May 12. PMID 32407786
- [Result] Leblebicioglu H, Erben N, Rosenthal VD, Sener A, Uzun C, Senol G, Ersoz G, Demirdal T, Duygu F, Willke A, Sirmatel F, Oztoprak N, Koksal I, Oncul O, Gurbuz Y, Guclu E, Turgut H, Yalcin AN, Ozdemir D, Kendirli T, Aslan T, Esen S, Ulger F, Dilek A, Yilmaz H, Sunbul M, Ozgunes I, Usluer G, Otkun M, Kaya A, Kuyucu N, Kaya Z, Meric M, Azak E, Yylmaz G, Kaya S, Ulusoy H, Haznedaroglu T, Gorenek L, Acar A, Tutuncu E, Karabay O, Kaya G, Sacar S, Sungurtekin H, Ugurcan D, Turhan O, Kaya S, Gumus E, Dursun O, Geyik MF, Sahin A, Erdogan S, Ince E, Karbuz A, Ciftci E, Tasyapar N, Gunes M. Surgical site infection rates in 16 cities in Turkey: findings of the International Nosocomial Infection Control Consortium (INICC). Am J Infect Control. 2015 Jan;43(1):48-52. doi: 10.1016/j.ajic.2014.09.017. PMID 25564124
- [Result] Ruhstaller K, Downes KL, Chandrasekaran S, Srinivas S, Durnwald C. Prophylactic Wound Vacuum Therapy after Cesarean Section to Prevent Wound Complications in the Obese Population: A Randomized Controlled Trial (the ProVac Study). Am J Perinatol. 2017 Sep;34(11):1125-1130. doi: 10.1055/s-0037-1604161. Epub 2017 Jul 13. PMID 28704847
- [Result] Hadiati DR, Hakimi M, Nurdiati DS, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2018 Oct 22;10(10):CD007462. doi: 10.1002/14651858.CD007462.pub4. PMID 30346040
- [Result] Ngai IM, Van Arsdale A, Govindappagari S, Judge NE, Neto NK, Bernstein J, Bernstein PS, Garry DJ. Skin Preparation for Prevention of Surgical Site Infection After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2015 Dec;126(6):1251-1257. doi: 10.1097/AOG.0000000000001118. PMID 26551196
- [Result] Kunkle CM, Marchan J, Safadi S, Whitman S, Chmait RH. Chlorhexidine gluconate versus povidone iodine at cesarean delivery: a randomized controlled trial. J Matern Fetal Neonatal Med. 2015 Mar;28(5):573-7. doi: 10.3109/14767058.2014.926884. Epub 2014 Jun 18. PMID 24849000
- [Result] Sahin S, Sinan O. Investigation of mothers' postpartum breastfeeding and comfort conditions. Health Care Women Int. 2021;42(4-6):913-924. doi: 10.1080/07399332.2021.1883022. Epub 2021 Mar 8. PMID 33683176
- [Result] Zengin H, Bafali IO, Caka SY, Tiryaki O, Cinar N. Childbirth and Postpartum Period Fear and the Related Factors in Pregnancy. J Coll Physicians Surg Pak. 2020 Feb;30(2):144-148. doi: 10.29271/jcpsp.2020.02.144. PMID 32036820
- [Result] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Result] Brown CR, Dodds L, Legge A, Bryanton J, Semenic S. Factors influencing the reasons why mothers stop breastfeeding. Can J Public Health. 2014 May 9;105(3):e179-85. doi: 10.17269/cjph.105.4244. PMID 25165836
- [Result] Edmiston CE Jr, Bruden B, Rucinski MC, Henen C, Graham MB, Lewis BL. Reducing the risk of surgical site infections: does chlorhexidine gluconate provide a risk reduction benefit? Am J Infect Control. 2013 May;41(5 Suppl):S49-55. doi: 10.1016/j.ajic.2012.10.030. PMID 23622749
- [Result] Kapadia BH, Johnson AJ, Daley JA, Issa K, Mont MA. Pre-admission cutaneous chlorhexidine preparation reduces surgical site infections in total hip arthroplasty. J Arthroplasty. 2013 Mar;28(3):490-3. doi: 10.1016/j.arth.2012.07.015. Epub 2012 Oct 29. PMID 23114192
- [Result] Jakobsson J, Perlkvist A, Wann-Hansson C. Searching for evidence regarding using preoperative disinfection showers to prevent surgical site infections: a systematic review. Worldviews Evid Based Nurs. 2011 Sep;8(3):143-52. doi: 10.1111/j.1741-6787.2010.00201.x. Epub 2010 Sep 28. PMID 20880006
- [Result] Karki S, Cheng AC. Impact of non-rinse skin cleansing with chlorhexidine gluconate on prevention of healthcare-associated infections and colonization with multi-resistant organisms: a systematic review. J Hosp Infect. 2012 Oct;82(2):71-84. doi: 10.1016/j.jhin.2012.07.005. Epub 2012 Aug 11. PMID 22889522
- [Result] Barreto R, Barrois B, Lambert J, Malhotra-Kumar S, Santos-Fernandes V, Monstrey S. Addressing the challenges in antisepsis: focus on povidone iodine. Int J Antimicrob Agents. 2020 Sep;56(3):106064. doi: 10.1016/j.ijantimicag.2020.106064. Epub 2020 Jun 26. PMID 32599228
- [Result] Haas DM, Morgan S, Contreras K, Enders S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2018 Jul 17;7(7):CD007892. doi: 10.1002/14651858.CD007892.pub6. PMID 30016540
- [Result] Dumville JC, McFarlane E, Edwards P, Lipp A, Holmes A. Preoperative skin antiseptics for preventing surgical wound infections after clean surgery. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003949. doi: 10.1002/14651858.CD003949.pub3. PMID 23543526
- [Result] Tuuli MG, Liu J, Stout MJ, Martin S, Cahill AG, Odibo AO, Colditz GA, Macones GA. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. N Engl J Med. 2016 Feb 18;374(7):647-55. doi: 10.1056/NEJMoa1511048. Epub 2016 Feb 4. PMID 26844840
- [Result] Chlebicki MP, Safdar N, O'Horo JC, Maki DG. Preoperative chlorhexidine shower or bath for prevention of surgical site infection: a meta-analysis. Am J Infect Control. 2013 Feb;41(2):167-73. doi: 10.1016/j.ajic.2012.02.014. Epub 2012 Jun 19. PMID 22722008
- [Result] Kasai KE, Nomura RM, Benute GR, de Lucia MC, Zugaib M. Women's opinions about mode of birth in Brazil: a qualitative study in a public teaching hospital. Midwifery. 2010 Jun;26(3):319-26. doi: 10.1016/j.midw.2008.08.001. Epub 2008 Oct 7. PMID 18842327
- See also: Centers for Disease Control and Prevention. (2021). Births: Final data for 2019 — https://www.cdc.gov/nchs/data/nvsr/nvsr70/nvsr70-02-508.
- See also: Turkish Society of Gynecology and Obstetrics, Ministry of Health — https://www.tjod.org/saglik-bakanligi-tjod-sezaryen-oranlarini-azaltma-ortak-eylem-plani/